CLINICAL TRIAL: NCT02685787
Title: Can Early Counseling and Support for Alzheimer's Disease Caregivers Improve Burden? A Multi-centre Active Randomized Clinical Trial in Local Health Services
Brief Title: Early Counseling and Support for Alzheimer's Disease Caregivers
Acronym: D_CareGiver
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria Locale N.1 dell'Umbria (Other)
Collaborators: Azienda Ospedaliera di Perugia (Other); Azienda Ospedaliera di Terni (Unknown); Azienda Unità Sanitaria Locale Umbria n. 2 (Unknown)
Responsible Party: Principal Investigator, Serena Amici, MD, Azienda Sanitaria Locale N.1 dell'Umbria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR-2009-1607340
Record Dates: First submitted 2016-02-06; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Alzheimer's Disease
Keywords: Care-giver burden; Dementia; Alzheimer's disease; Care-giver depression; Care-giver anxiety
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychosocial Intervention (Experimental): Every caregiver in this arm will be assigned to a permanent counselor.
  Interventions: Behavioral: Psychosocial Intervention
- Educational Intervention on AD (Active Comparator): The caregiver enrolled in this arm will not be assigned to a counselor but will participate to group sessions on AD education.
  Interventions: Behavioral: Educational Intervention on AD

INTERVENTIONS:
Behavioral: Psychosocial Intervention — The caregiver in the intervention arm will meet the counselors six times. The first and the last sessions will be attended by the caregiver only whereas the remaining four sessions will be attended by the caregiver and other family members. Interventions will be tailored for the caregivers based upon: 1) depression and anxiety; 2) burden; 3) self care and health-related behavior; 4) social support; and 5) behavioral symptoms. The design and management of the structured intervention will follow a published counseling caregiver manual, based on the experiences matured at New York University. Every session will be documented.
  Arms: Psychosocial Intervention
Behavioral: Educational Intervention on AD — The caregiver enrolled in this arm:1) will not receive counseling or support; 2) will participate to group sessions; 3) the six hours sessions will divulge information on AD using a slide-show. Each session will focus on the following topic: (a) diagnosis and treatment b) cognitive deficit management, c) behavioral disturbance management, d) daily living management, e) non-pharmacological treatment, f) legal issues and available health and social services.
  Additionally, contrary to other arm, caregivers will not receive any telephone calls after the end of the educational sessions.
  Arms: Educational Intervention on AD

SUMMARY:
This randomized trial evaluates the efficacy of counselling for reducing anxiety and depression in caregivers of patients with dementia. Half of the participants will receive six hours providing counselling and psycho-social support to caregivers along with a specific telephone support service - Ad Hoc Telephone Counselling whereas the remaining participants will receive six hours providing general information about Alzheimer Disease.

DETAILED DESCRIPTION:
This study will be a multicentre Umbrian PROBE design (treatment regimens are blinded to both caregivers and evaluators) with investigating the effectiveness comparing two active treatment "counseling and support" versus "educational group focusing on AD" in 230 primary caregivers of AD patients.

If all inclusion criteria are met, the caregiver will be asked to sign a written informed consent form. Failure to do so, will result in exclusion from the study. The treatment will not be disclosed to the caregivers, although the caregivers will be told that they will participate in a study with two different active treatments which will require a total of six-hour sessions.

Care providers and Study settings

Caregiver will be recruited in secondary outpatient clinic located in Umbrian health maintenance organizations (HMO). Outpatient clinic in Umbria are disseminated in the territory and each small city has its own clinic (Città di Castello, Foligno, Gualdo Tadino, Gubbio, Perugia, Marsciano, Passignano, San Giustino, Spoleto, Terni, Todi, Umbertide with population ranging from 11,000 to 166,000 inhabitants, of them around 70% living in the country/small village). Care providers were neurologist and geriatrician with twelve to 30 year experience in dementia practice, working in high volume outpatient clinic.

INTERVENTION

Treatment arm

Psychosocial Intervention

Every caregiver will be assigned to a permanent counselor. The caregiver in the intervention arm will meet the counselors six times in person. The first and the last sessions will be attended by the caregiver only whereas the remaining four sessions will be attended by the caregiver and other family members who are involved in the daily management of the patient. All meetings will held within 4 months of the initial assessment. Interventions will be tailored for the caregivers based upon:

1. depression and anxiety;
2. burden;
3. self care and health-related behavior;
4. social support; and
5. behavioral symptoms.

The design and management of the structured intervention will follow a published counseling caregiver manual, based on the experiences matured at New York University. Every session will be documented.

Moreover, the counselor will make three ad hoc telephone calls to the caregiver each month following the six in-person sessions counseling, in order to monitor the well-being of the caregiver. Telephone communications will be documented; other types of communication will not be considered valid (e.g. telephone text messages or social network messages).

Finally, the counselor will be available to the caregiver via a telephone service.

All counselors will meet monthly to update the the adherence to the protocol to resolve any problems.

Educational Intervention on AD

The caregiver enrolled in this arm:

1. will not receive counseling or support;
2. will participate to group sessions;
3. the six hours sessions will divulge information on AD using a slide-show.

Each session will focus on the following topic:

1. diagnosis and treatment,
2. cognitive deficit management,
3. behavioral disturbance management,
4. daily living management,
5. non-pharmacological treatment,
6. legal issues and available health and social services.

Additionally, contrary to other arm, caregivers will not receive any telephone calls after the end of the educational sessions.

Whenever a caregiver in this arm requires additional support, he/she will be referred to volunteers of the local Alzheimer's Association.

Follow-up evaluation

Caregivers will be evaluated at 6, 12, and 24 months after baseline evaluation; outcome measures will repeated at every evaluation. Patients will be evaluated every twelve months after baseline, as standard care requires. The implementation of the intervention program will be closely monitored, including activities as well as outcomes. The activities and progress of each caregiver and family will be tracked. The participation and attrition rate will be calculated and reported; the causes of delays in scheduling or attrition due to a move to another city or state, hospitalization, a nursing home admission, or death will be recorded.

The study will be under constant monitoring of an External Committee.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver actively caring the patient for at least 4 hours a day over the last 6 months.
* Their patients must have scored lower than 24 on the Mini-Mental State Examination score, at screening.
* Their patients must have at least one limitation according to the Activities of Daily Living (ADL) test, or two limitations based on the Instrumental Activities of Daily Living (IADL) test.

Exclusion Criteria:

* Self-reported current psychiatric history, not related to patient's disease
* caregiver of non-AD dementias
* their patients could not undergo clinical and neuropsychological evaluation
* caregiver with insufficient Italian language knowledge
* can not be contacted by telephone regularly (eg. Do not have telephone/mobile, severe auditory deficits).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2012-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Care-giver burden measured with Zarit Burden Inventory (ZBI) | ZBI evaluated at 6 months
  Change from baseline of care-giver burden at 6 months
Care-giver burden measured with ZBI | ZBI evaluated at 12 months
  Change from baseline of care-giver burden at 12 months
Care-giver burden measured with ZBI | ZBI evaluated at 24 months
  Change from baseline of care-giver burden at 24 months

SECONDARY OUTCOMES:
Caregiver depression measured using the Hospital Anxiety and Depression Scale (HADS) | At baseline, and after 6 months, 12 and 24 months from baseline
Behavioural and psychological symptoms of dementia (BPSD) using the Neuropsychiatric Inventory (NPI) | At baseline, and after 6 months, 12 and 24 months from baseline
BPSD using the Revised Memory and Behaviour Checklist (RMBC) | At baseline, and after 6 months, 12 and 24 months from baseline
Patient quality-of-life measure with Logdson's Quality of Life AD | At baseline, and after 6 months, 12 and 24 months from baseline
Care-giver quality-of-life measure with Euro-Quality of Life | At baseline, and after 6 months, 12 and 24 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Montedori, MD, Study Chair — Regional Health Authority of Umbria
Locations (1):
- USL Umbria 1, Perugia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Adelman RD, Tmanova LL, Delgado D, Dion S, Lachs MS. Caregiver burden: a clinical review. JAMA. 2014 Mar 12;311(10):1052-60. doi: 10.1001/jama.2014.304. PMID 24618967
- [Result] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Result] Andren S, Elmstahl S. Effective psychosocial intervention for family caregivers lengthens time elapsed before nursing home placement of individuals with dementia: a five-year follow-up study. Int Psychogeriatr. 2008 Dec;20(6):1177-92. doi: 10.1017/S1041610208007503. Epub 2008 Jul 8. PMID 18606052
- [Result] Binetti G, Mega MS, Magni E, Padovani A, Rozzini L, Bianchetti A, Trabucchi M, Cummings JL. Behavioral disorders in Alzheimer disease: a transcultural perspective. Arch Neurol. 1998 Apr;55(4):539-44. doi: 10.1001/archneur.55.4.539. PMID 9561983
- [Result] Brodaty H, Green A, Koschera A. Meta-analysis of psychosocial interventions for caregivers of people with dementia. J Am Geriatr Soc. 2003 May;51(5):657-64. doi: 10.1034/j.1600-0579.2003.00210.x. PMID 12752841
- [Result] Chattat R, Cortesi V, Izzicupo F, Del Re ML, Sgarbi C, Fabbo A, Bergonzini E. The Italian version of the Zarit Burden interview: a validation study. Int Psychogeriatr. 2011 Jun;23(5):797-805. doi: 10.1017/S1041610210002218. Epub 2010 Dec 16. PMID 21205379
- [Result] Cuijpers P. Depressive disorders in caregivers of dementia patients: a systematic review. Aging Ment Health. 2005 Jul;9(4):325-30. doi: 10.1080/13607860500090078. PMID 16019288
- [Result] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Result] Joling KJ, van Marwijk HW, Smit F, van der Horst HE, Scheltens P, van de Ven PM, Mittelman MS, van Hout HP. Does a family meetings intervention prevent depression and anxiety in family caregivers of dementia patients? A randomized trial. PLoS One. 2012;7(1):e30936. doi: 10.1371/journal.pone.0030936. Epub 2012 Jan 27. PMID 22303473
- [Result] Mittelman MS, Brodaty H, Wallen AS, Burns A. A three-country randomized controlled trial of a psychosocial intervention for caregivers combined with pharmacological treatment for patients with Alzheimer disease: effects on caregiver depression. Am J Geriatr Psychiatry. 2008 Nov;16(11):893-904. doi: 10.1097/JGP.0b013e3181898095. PMID 18978250
- [Result] Mittelman MS, Haley WE, Clay OJ, Roth DL. Improving caregiver well-being delays nursing home placement of patients with Alzheimer disease. Neurology. 2006 Nov 14;67(9):1592-9. doi: 10.1212/01.wnl.0000242727.81172.91. PMID 17101889
- [Result] Schulz R, Beach SR. Caregiving as a risk factor for mortality: the Caregiver Health Effects Study. JAMA. 1999 Dec 15;282(23):2215-9. doi: 10.1001/jama.282.23.2215. PMID 10605972
- [Result] Schulz R, Martire LM. Family caregiving of persons with dementia: prevalence, health effects, and support strategies. Am J Geriatr Psychiatry. 2004 May-Jun;12(3):240-9. PMID 15126224
- [Result] Wimo A, Jonsson L, Zbrozek A. The Resource Utilization in Dementia (RUD) instrument is valid for assessing informal care time in community-living patients with dementia. J Nutr Health Aging. 2010 Oct;14(8):685-90. doi: 10.1007/s12603-010-0316-2. PMID 20922346